CLINICAL TRIAL: NCT04113356
Title: Clinical Relevance of Magnetic Resonance Imaging in Acute ST-Elevation Myocardial Infarction
Brief Title: Magnetic Resonance Imaging In Acute ST-Elevation Myocardial Infarction
Acronym: MARINA-STEMI
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: AN3775
Record Dates: First submitted 2019-08-23; First posted 2019-10-02 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Acute ST-Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ST-Elevation Myocardial Infarction: Patients with acute ST-elevation myocardial infarction treated with primary percutaneous coronary intervention
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance Imaging — Cardiovascular magnetic resonance imaging will be performed within the first week after ST-elevation myocardial infarction and in a defined subgroup 4 months, 12 months and 10 years thereafter.

SUMMARY:
Cardiovascular magnetic resonance imaging enables comprehensive assessment of cardiovascular function, morphology and pathology. The investigators aim to evaluate the nature and clinical significance of magnetic resonance imaging parameters in patients presenting with first acute ST-elevation myocardial infarction.

ELIGIBILITY:
Inclusion criteria:

* First ST-elevation myocardial infarction according to the European Society of Cardiology/American College of Cardiology committee criteria
* Primary percutaneous coronary intervention within 24 hours after symptom onset

Exclusion criteria:

* Age < 18 years
* Any history of a previous myocardial infarction or coronary intervention
* Clinically unstable patients (Killip class >2)
* Renal failure (estimated glomerular filtration rate < 30 ml/min/1.73 m2)
* Contraindications to cardiac magnetic resonance imaging (pacemaker, cerebral aneurysm clip, orbital foreign body, known or suggested contrast allergy to gadolinium, claustrophobia)
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ST-elevation myocardial infarction treated with primary percutaneous coronary intervention admitted to the coronary care unit of Innsbruck University Hospital for Internal Medicine III (Cardiology and Angiology).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Occurence of major adverse cardiovascular events | 1 - 5 years

SECONDARY OUTCOMES:
Infarct size assessment (% of left ventricular myocardial mass) | baseline, 4 months and 12 months
Assessment of infarct transmurality grade (%) with late gadolinium enhancement imaging | baseline, 4 months and 12 months
Occurence and area of microvascular obstruction | baseline
Intramyocardial haemorrhage assessed by T2* imaging | baseline, 4 months and 12 months
Tissue characterisation by T1, T2 and T2* Mapping | baseline, 4 months and 12 months
Myocardial deformation by strain analysis | baseline, 4 months and 12 months
Chamber volumes by cine imaging | baseline, 4 months and 12 months
Cardiac function by cine imaging | baseline, 4 months and 12 months
Stroke volumes by phase contrast imaging | baseline, 4 months and 12 months
Aortic pulse wave velocity and distensibility by phase contrast imaging | baseline, 4 months and 12 months
Aortic pulse wave distensibility by phase contrast imaging | baseline, 4 months and 12 months
Quality of life and invalidity assessment (Global Physical Activity Questionnaire) | 1 - 5 years
Biomarker release during the acute and subacute phase | baseline, 4 months and 12 months
  biomarker concentrations of hemodynamic stress (n-terminal pro-B-type natriuretic peptide), neurohumoral markers (i.e. neprilysin ng/ml), inflammatory markers (i.e. procalcitonin µg/l) and markers of myocardial injury (i.e. high sensitivity cardiac troponin T ng/l)
Parameters of cardiac function by transthoracic echocardiography | baseline, 4 months and 12 months
Plaque volume by 3D ultrasound | baseline, 12 months
Cardiac autonomic function | baseline, 4 months and 12 months
  Deceleration capacity of heart rate
Cardiac autonomic function | baseline, 4 months and 12 months
  Heart rate variability
Cardiac autonomic function | baseline, 4 months and 12 months
  Periodic repolarization dynamics
Cardiac autonomic function | baseline, 4 months and 12 months
  Baroreflex sensitivity
Cardiac autonomic function | baseline, 4 months and 12 months
  Skin sympathetic nerve activity

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Metzler, MD, MSc, Principal Investigator — University Hospital for Internal Medicine III (Cardiology and Angiology)
Locations (2):
- Austria (2):
  - University Hospital for Internal Medicine III (Cardiology and Angiology), Innsbruck
  - University Hospital for Radiology, Innsbruck

REFERENCES:
- [Derived] Lechner I, Reindl M, von der Emde S, Desheva A, Oberhollenzer F, Tiller C, Holzknecht M, Kremser T, Faccini J, Gollmann-Tepekoylu C, Kremser C, Mayr A, Bauer A, Metzler B, Reinstadler SJ. Hepatic Tissue Alterations in ST-Elevation Myocardial Infarction: Determinants and Prognostic Implications. Circ Cardiovasc Imaging. 2024 Dec;17(12):e017041. doi: 10.1161/CIRCIMAGING.124.017041. Epub 2024 Nov 29. PMID 39611252
- [Derived] Tiller C, Holzknecht M, Lechner I, Oberhollenzer F, von der Emde S, Kremser T, Gollmann-Tepekoylu C, Mayr A, Bauer A, Metzler B, Reinstadler SJ, Reindl M. Association of Circulating PCSK9 With Ischemia-Reperfusion Injury in Acute ST-Elevation Myocardial Infarction. Circ Cardiovasc Imaging. 2024 Aug;17(8):e016482. doi: 10.1161/CIRCIMAGING.123.016482. Epub 2024 Aug 20. PMID 39163371
- [Derived] Holzknecht M, Tiller C, Reindl M, Lechner I, Fink P, Lunger P, Mayr A, Henninger B, Brenner C, Klug G, Bauer A, Metzler B, Reinstadler SJ. Association of C-Reactive Protein Velocity with Early Left Ventricular Dysfunction in Patients with First ST-Elevation Myocardial Infarction. J Clin Med. 2021 Nov 24;10(23):5494. doi: 10.3390/jcm10235494. PMID 34884196
- [Derived] Tiller C, Reindl M, Holzknecht M, Lechner I, Schwaiger J, Brenner C, Mayr A, Klug G, Bauer A, Metzler B, Reinstadler SJ. Association of plasma interleukin-6 with infarct size, reperfusion injury, and adverse remodelling after ST-elevation myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2022 Feb 8;11(2):113-123. doi: 10.1093/ehjacc/zuab110. PMID 34849677
- [Derived] Lechner I, Reindl M, Tiller C, Holzknecht M, Niederreiter S, Mayr A, Klug G, Brenner C, Bauer A, Metzler B, Reinstadler SJ. Determinants and prognostic relevance of aortic stiffness in patients with recent ST-elevation myocardial infarction. Int J Cardiovasc Imaging. 2022 Jan;38(1):237-247. doi: 10.1007/s10554-021-02383-0. Epub 2021 Sep 2. PMID 34476665
- [Derived] Reindl M, Lechner I, Tiller C, Holzknecht M, Rangger A, Mayr A, Theurl M, Klug G, Brenner C, Bauer A, Metzler B, Reinstadler SJ. Glycemic Status and Reperfusion Injury in Patients With ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Imaging. 2021 Sep;14(9):1875-1877. doi: 10.1016/j.jcmg.2021.04.007. Epub 2021 May 19. No abstract available. PMID 34023265
- [Derived] Reindl M, Tiller C, Holzknecht M, Lechner I, Eisner D, Riepl L, Pamminger M, Henninger B, Mayr A, Schwaiger JP, Klug G, Bauer A, Metzler B, Reinstadler SJ. Global longitudinal strain by feature tracking for optimized prediction of adverse remodeling after ST-elevation myocardial infarction. Clin Res Cardiol. 2021 Jan;110(1):61-71. doi: 10.1007/s00392-020-01649-2. Epub 2020 Apr 15. PMID 32296969